CLINICAL TRIAL: NCT01800097
Title: Treatment of Post Stroke Fatigue With Modafinil, Effect on Rehabilitation, Fatigue and Bonemass Index
Brief Title: Treatment of Post Stroke Fatigue With a Wakefulness Promoting Agent
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Karsten Overgaard, Principal Investigator, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ModaA001
Record Dates: First submitted 2012-10-23; First posted 2013-02-27 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Stroke; Post Stroke Fatigue
Keywords: stroke; fatigue; modafinil
MeSH Terms: conditions — Stroke; Fatigue | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo
- Modafinil (Active Comparator): Modafinil
  Interventions: Drug: modafinil

INTERVENTIONS:
Drug: modafinil — Tablet, 400 mg once daily, morning (200 mg if age 65 or above) for 3 months
  Other Names: modiodal, provigil
  Arms: Modafinil
Drug: placebo — Tablets, 400 mg once daily ( 200 mg if age 65 or above)morning for 3 months.
  Arms: placebo

SUMMARY:
This study is an investigator initiated placebo controlled double blinded trial. The hypothesis is that treatment with modafinil positively will affect behavioural and cognitive rehabilitation after stroke, causing the treatment group to experience decreased fatigue, increased endurance, improved skills of sustaining attention and faster reaction times. The cognitive rehabilitation will show in increased muscle mass, decreased osteoporosis and better physical performances due to a higher level of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and stroke within 14 days
* Modified Rankin Scale 3 or under and Barthel 85 or over before stroke
* Person that can understand instruction and do tests and questionnaires on their own or with support
* has given informed consent
* MFI-20 score of 12 or more
* Infertile person or fertile women tested negative of pregnancy and using safe anticonception

Exclusion Criteria:

* Dementia or other neuropsychiatric disease making the person incapable of understanding instructions
* Other disease with fatigue as a known symptom
* stroke induced by trauma, infection or surgical procedure
* former drug abuse
* known contraindication to treatment with modafinil
* known active malignancy, benign intracranial tumor, subdural or epidural bleeding
* kidneydysfunction with creatinin more than 265 micromol/L or liver disease with ASAT (aspartate aminotransferase) elevated to more than 70 U/L for women or 100 U/L for men.
* allergy to project treatment
* use of benzodiazepin or antiepileptic drugs in a fixed dose. Sleeping pills not included.
* Patients threaded with ciclosporin or anti HIV medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Multidimensional Fatigue Inventory (MFI- 20) | 3 months
  Questionnaire

SECONDARY OUTCOMES:
MFI-20 | 1 month
  Questionnaire
MFI-20 | 6 months
  Questionnaire
Fatigue severity scale (FSS) | 3 months
FSS | 1 month
  Questionnaire
FSS | 6 months
  Questionnaire

OTHER OUTCOMES:
Change in bone mineral density and musclemass from baseline to 3 months | 3 months
  DXA-scans. (dual energy x-ray absorptiometry)
Reactiontime | 1 month
  A special designed computerprogramme will be used to measure the patients reactiontime.
Stroke Specific Quality Of Life (SSQOL) | 3 months
  Questionnaire
Change in Barthel Index | 3 months
  score
Modified Ranking Scale | 3 months
  score
Multidimensional Depression Inventory | 3 months
  Questionnaire
Change in "Time up and go" and "chair to stand test" from baseline | 3 months
Cognitive performance, Montreal Cognitive Assessment(MOCA) | 3 months
  test
Change in bone mineral density and musclemass from baseline to 6 months | 6 months
  DXA-scan
Reactiontime | 3 months
  A special designed computerprogramme will be used to measure the patients reactiontime.
Reactiontime | 6 months
  A special designed computerprogramme will be used to measure the patients reactiontime.
Stroke Specific Quality Of Life | 6 months
  Questionnaire
Change in Barthel Index | 6 months
Modified Ranking Scale | 6 months
  score
Change in "Time up and go" and "chair to stand test" from baseline | 6 months
Multidimensional Depression Inventory | 6 months
  Questionnaire
Cognitive performance, Montreal Cognitive Assessment(MOCA) | 6 months
  test
Stroke Specific Quality Of Life (SSQOL) | 1 month
  Questionnaire
Change in Barthel Index | 1 month
  score
Modified Ranking Scale | 1 month
  score
Multidimensional Depression Inventory | 1 month
  Questionnaire
Change in "Time up and go" and "chair to stand test" from baseline | 1 month
Cognitive performance, Montreal Cognitive Assessment(MOCA) | 1 month
  test

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Overgaard, MD, Principal Investigator — Department of Neurology, Herlev Hospital
Locations (1):
- Department of Neurology, Herlev Hospital,, Herlev, Denmark

REFERENCES:
- [Derived] Poulsen MB, Damgaard B, Zerahn B, Overgaard K, Rasmussen RS. Modafinil May Alleviate Poststroke Fatigue: A Randomized, Placebo-Controlled, Double-Blinded Trial. Stroke. 2015 Dec;46(12):3470-7. doi: 10.1161/STROKEAHA.115.010860. Epub 2015 Nov 3. PMID 26534969